CLINICAL TRIAL: NCT05823805
Title: Approaches For ThE pRioritization of Patients in priMAry Care Post-COVID To Reduce Health Inequities (AFTERMATH): Cluster Randomized Controlled Trial
Brief Title: Approaches For ThE pRioritization of Patients in priMAry Care Post-COVID To Reduce Health Inequities (AFTERMATH)
Acronym: AFTERMATH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AFTERMATH
Record Dates: First submitted 2023-04-19; First posted 2023-04-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: primary health care; primary care; schizophrenia; bipolar disorder; cluster randomized controlled trial; community health worker; randomized controlled trial
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder | interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community Health Worker + Quality Improvement reports (Experimental): Family physicians with ten or more patients living with schizophrenia and/or bipolar disorder will work with a community health worker who will assist them in reviewing their individualized reports, which presents data on patient's preventive health care status and engagement in care.
  Interventions: Other: Community Health Worker
- Quality Improvement dashboard (No Intervention): Family physicians with ten or more patients living with schizophrenia and/or bipolar disorder will have access to an individualized reports, which presents data on patient's preventive health care status and engagement in care.

INTERVENTIONS:
Other: Community Health Worker — Physicians will work with a Community Health Worker (CHW) to review the data presented in their Quality Improvement reports, and triage patients for proactive outreach (e.g. "No action necessary", "Call patient to check-in", "Arrange BP, weight and labs", "Book for phone appointment", "Book for in-person appointment").
  Arms: Community Health Worker + Quality Improvement reports

SUMMARY:
The COVID-19 pandemic significantly impacted primary care across Canada. Inequities in prevention activities and chronic disease management likely increased but the extent is unknown. Pragmatic interventions are required to prioritize patients and improve the quality of primary care post-COVID. In AFTERMATH, the investigators will conduct a pragmatic cluster randomized controlled trial (cRCT) at the largest primary care Practice-Based Research Network (PBRN) in Ontario, focused on a highly marginalized population: adults living with mental illness and one or more additional chronic diseases. The investigators will test an intervention that builds on the investigators' past work and combines data and supports to primary care providers to improve quality of life, reduce gaps in prevention activities and improve chronic disease management. The investigators' project will result in new evidence on ways to improve access to care and reduce inequities, and inform future efforts to use data beyond COVID-19.

ELIGIBILITY:
Inclusion Criteria:

A. Family physicians: Any family physician in a University of Toronto DFCM academic site with 10+ community-dwelling patients living with schizophrenia or bipolar disorder plus one or more additional chronic disease (COPD, diabetes, hypertension, osteoarthritis, dementia, epilepsy and Parkinson's).

B. Patients: Patients from the included family physician practices living with schizophrenia or bipolar disorder plus one or more additional chronic disease (COPD, diabetes, hypertension, osteoarthritis, dementia, epilepsy and Parkinson's).

Exclusion Criteria:

A. Family Physicians: None

B. Patients: Patients under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
health-related quality of life | 9 months
  We will assess health-related quality of life using the World Health Organization WHO QOL-BREF scale

SECONDARY OUTCOMES:
Preventive care activities and chronic disease management outcomes | 9 months
  Preventive care activities up-to-date and chronic disease management outcomes, which reflect the goals of primary care teams, and health services outcomes (primary care visits, emergency department visits, hospitalizations, and total health services costs).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pinto, MD MSc, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be made available to qualified researchers with academic interest in primary care health equity research and mental health research. Data will only be made available to interested parties after all applicable agreements have been executed.
Time Frame: Requests to access the data can be made beginning 3 months and up until 2 years after article publication.
Access Criteria: Access to study IPD will be granted to qualified researchers upon approval of their Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). To submit a request or for any additional questions, please contact Upstreamlab@unityhealth.to.
URL: https://upstreamlab.org/project/aftermath/

REFERENCES:
- See also: AFTERMATH study website — https://upstreamlab.org/project/aftermath/